CLINICAL TRIAL: NCT00795366
Title: Vasopressin Versus Catecholamines for Cerebral Perfusion Pressure Control in Brain Injured Trauma Patients
Acronym: AVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Kenneth Proctor, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060949
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Traumatic Brain Injury
Keywords: TBI, trauma, brain
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries | interventions — Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AVP, arginine vasopressin (Active Comparator): Vasopressin
  Interventions: Drug: arginine vasopressin
- Standard Catecholamine (Active Comparator): levophed, dopamine, phenylephrine)
  Interventions: Drug: Standard catecholamine

INTERVENTIONS:
Drug: arginine vasopressin — Titrated to cerebral perfusion pressure greater than 60 mm Hg
  Arms: AVP, arginine vasopressin
Drug: Standard catecholamine — Titrated catecholamine of attending physicians preference to cerebral perfusion pressure greater than 60 mm Hg.
  Arms: Standard Catecholamine

SUMMARY:
Traumatic brain injury (TBI) is among the leading causes of trauma death and disability in both civilian and military populations. The damage that occurs at the instant of trauma cannot be modified; the secondary injuries that occur afterward are the impediments to recovery and can be influenced by the physician. Cerebral ischemia is the most important secondary event that determines outcome following TBI. To minimize ischemic episodes once the patient has arrived at the hospital, most treatments are aimed at optimizing cerebral perfusion pressure (CPP). The cornerstones of these treatments include mannitol, to reduce intracranial pressure (ICP), and catecholamines, such as phenylephrine (PE), to increase mean arterial pressure (MAP), but these agents have undesired side effects. Nevertheless, once they lose potency, there are few alternatives. The main objective of this proposal to develop a new therapeutic option for CPP management in TBI patients using arginine vasopressin (AVP).

AVP is the endogenous anti-diuretic hormone. It is FDA-approved for use in the diagnosis and treatment of diabetes insipidus, for the prevention and treatment of post-operative abdominal distention, and in abdominal radiography to dispel interfering gas shadows. It has been used off-label for several other conditions. There is minimal information on its therapeutic potential after TBI. The investigators have demonstrated that AVP during fluid resuscitation rapidly restored hemodynamics, CPP, and improves acute survival in a clinically-relevant model of TBI. The investigators observed similar short term benefits after chest and liver trauma. Nevertheless, AVP has actions that could mask any short term benefit. The investigators have already defined risks and benefits of AVP therapy, relative to PE, in four different clinically-relevant laboratory model. The investigators now plan to evaluate this new therapy relative to the current evidence-based guideline for CPP management in TBI patients.

The working hypothesis is that the risk/benefit profile for AVP is equal, or superior to, PE at equi-effective doses for the management of CPP following TBI. A corollary is that a higher CPP can be safely tolerated with AVP vs catecholamines.

THE INVESTIGATORS AIM TO: Determine whether AVP is safe and effective to maintain CPP = 60 mm Hg in TBI patients.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label clinical trial comparing vasopressin and catecholamines for cerebral perfusion pressure (CPP) control after a traumatic brain injury (TBI).

Once a neurosurgeon is consulted for a patient presenting with a TBI, they will review entry criteria and refer to study personnel to obtain informed consent.

After informed consent, subjects will be randomized into one of the 2 groups to receive either a catecholamine at the discretion of the attending physicians or vasopressin (AVP). A 6 hour dose of non-study drug will be permitted prior to initiation of study drug. The amount of study drug will be titrated to maintain cerebral perfusion pressure within normal limits. Subjects will be followed until they can maintain their CPP without vasopressor medication. Data collection will include amount and duration of vasopressor therapy and resulting cerebral perfusion pressure and time until successful weaning from vasopressor therapy.

All subsequent clinical care will be at the discretion of the attending physician.

The standard protocol/procedure for the discontinuation of drugs in each arm of the study is as follows: Vasopressors are discontinued in a step-wise fashion, regardless of the specific agent or the specific ICU patient population. In patients with severe traumatic brain injury (TBI), cerebral perfusion pressure (CPP) is maintained between 60 and 70 mmHg with vasopressors. When intracranial pressure (ICP) begins to correct (decrease), vasopressors are titrated downward slowly to maintain CPP. This continues until ICP is normalized and systemic hemodynamics are able to support a normal CPP. At this point, vasopressors are withdrawn completely. This process is standard regardless of the choice of vasopressor.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 yrs,
* Primary admission to the hospital within 8 h after injury
* Closed head injury
* Potential for intracranial pressure monitoring

Exclusion Criteria:

* Pregnant or nursing women
* Hemodynamic instability after initial resuscitation
* Vasopressor therapy for greater than 6 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Proctor, PhD, Principal Investigator — University of Miami
Locations (1):
- Ryder Trauma Center, Miami, Florida, United States

REFERENCES:
- [Background] Dudkiewicz M, Proctor KG. Tissue oxygenation during management of cerebral perfusion pressure with phenylephrine or vasopressin. Crit Care Med. 2008 Sep;36(9):2641-50. doi: 10.1097/CCM.0b013e3181847af3. PMID 18679110
- [Background] Sanui M, King DR, Feinstein AJ, Varon AJ, Cohn SM, Proctor KG. Effects of arginine vasopressin during resuscitation from hemorrhagic hypotension after traumatic brain injury. Crit Care Med. 2006 Feb;34(2):433-8. doi: 10.1097/01.ccm.0000196206.83534.39. PMID 16424725
- [Background] Feinstein AJ, Cohn SM, King DR, Sanui M, Proctor KG. Early vasopressin improves short-term survival after pulmonary contusion. J Trauma. 2005 Oct;59(4):876-82; discussion 882-3. doi: 10.1097/01.ta.0000187654.24146.22. PMID 16374276
- [Background] Feinstein AJ, Patel MB, Sanui M, Cohn SM, Majetschak M, Proctor KG. Resuscitation with pressors after traumatic brain injury. J Am Coll Surg. 2005 Oct;201(4):536-45. doi: 10.1016/j.jamcollsurg.2005.05.031. PMID 16183491

RESULTS

PARTICIPANT FLOW:
Groups:
- AVP, Arginine Vasopressin: Vasopressin: Titrated to cerebral perfusion pressure greater than 60 mm Hg
Period: Overall Study
Arm/Group | AVP, Arginine Vasopressin | Standard Catecholamine
Started | 42 | 54
Completed | 42 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AVP, Arginine Vasopressin: Vasopressin, arginine vasopressin: Titrated to cerebral perfusion pressure greater than 60 mm Hg
- Total: Total of all reporting groups
Arm/Group | AVP, Arginine Vasopressin | Standard Catecholamine | Total
Number analyzed (Participants) | 42 | 54 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (16) | 38 (18) | 39 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 34 | 43 | 77
Region of Enrollment [Number; unit: participants]
  United States | 42 | 54 | 96
ISS (Injury Severity Score) [Mean (Standard Deviation); unit: units on a scale] — ISS is an anatomical scoring system that provides an overall score for patients with multiple injuries. Each injury is assigned an Abbreviated Injury Scale (AIS) score and is allocated to one of six body regions (Head, Face, Chest, Abdomen, Extremities (including Pelvis), External). Only the highest AIS score in each body region is used. The 3 most severely injured body regions have their score squared and added together to produce the ISS score. The ISS scores range from 1 to 75, being one the least severe and 75 the most severe trauma injury.
  units on a scale | 29 (9) | 28 (10) | 28 (10)

OUTCOME MEASURES:

1. Primary Outcome: Time ICP >20
Description: The number of hours that participants remained with intracranial pressure above 20 mmHg
Time Frame: The number of hours during the first 5 days of intracranial pressure monitoring
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | AVP, Arginine Vasopressin | Standard Catecholamine
Number analyzed (Participants) | 42 | 54
Hours | 1.7 (1.8) | .9 (2.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the primary study period as the first 5 days of intracranial pressure monitoring while outcome data was also collected from admission until discharge from the hospital.
Arm/Group | AVP, Arginine Vasopressin | Standard Catecholamine
Serious Adverse Events (participants affected / at risk) | 6/42 | 6/54
Other Adverse Events (participants affected / at risk) | 0/42 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVP, Arginine Vasopressin (N=42) | Standard Catecholamine (N=54)
Death (General disorders) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No